CLINICAL TRIAL: NCT02601898
Title: Vaginal Administration of Alpha Lipoic Acid vs Progesterone for the Subchorionic Hematoma Treatment
Brief Title: Vaginal Administration of ALA vs Progesterone for the Subchorionic Hematoma Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Azienda USL Ferrara (Other Government)
Responsible Party: Principal Investigator, Demetrio Costantino, Medical Doctor, Azienda USL Ferrara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALAvsPROG
Record Dates: First submitted 2015-11-06; First posted 2015-11-11 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Subchorionic Hematoma in the First Trimester Pregnancy; Miscarriage
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Progesterone

ARMS (2):
- Lipoic acid (Experimental): vaginal capsules of lipoic acid (10 mg, one capsule per day)
  Interventions: Device: Lipoic acid
- Progesterone (Active Comparator): Vaginal soft gel of progesterone (200 mg, two capsules per day)
  Interventions: Drug: Progesterone

INTERVENTIONS:
Device: Lipoic acid — Vaginal capsules (medical device) containing 10 mg of lipoic acid (1 per day)
  Arms: Lipoic acid
Drug: Progesterone — Vaginal capsules (drug) containing 200 mg of progesterone (2 per day)
  Arms: Progesterone

SUMMARY:
The aim of this study was to compare the therapeutic efficacy of lipoic acid versus progesterone by vaginal administration on subchorionic hematoma resorption in women at the first trimester of pregnancy with threatened miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* Age: 24-37
* Gestational week: 7- 12
* Evidence of threatened miscarriage (pelvic pain with or without vaginal bleeding)
* Ultrasound evidence of subchorionic hematoma

Exclusion Criteria:

* Lack of fetus
* Absence of fetal heart tone
* Uterine anomaly or fetal anomaly
* Presence of multiple pregnancy
* Gestation pathology
* Therapies with anti-coagulants or anti-hypertensive drugs

Ages: 24 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in subchorionic hematoma from baseline at 20 days and 40 days, assessed as %improvement/worsening by ultrasoud examination | T1 (20 days); T2 (40 days)
  The evaluation of the hematoma significance is done comparing its size with that one of the gestational sac during the ultrasound examination. Changes in hematoma resorption (% improvement/ worsening) during the treatment were obtained for each patient by calculating the Δ percentage between two subsequent time points.

SECONDARY OUTCOMES:
Number of participants with abdominal pain as assessed by questionnaire | T1 (20 days)
Number of participants with vaginal bleeding as assessed by questionnaire | T1 (20 days)
Number of participants with abdominal pain as assessed by questionnaire | T2 (40 days)
  Questionaire
Number of participants with vaginal bleeding as assessed by questionnaire | T2 (40 days)
Number of participants who miscarried as assessed by ultrosound examination | 20 weeks of gestation

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda USL Ferrara, Ferrara, Italy

REFERENCES:
- [Background] Yassaee F, Shekarriz-Foumani R, Afsari S, Fallahian M. The effect of progesterone suppositories on threatened abortion: a randomized clinical trial. J Reprod Infertil. 2014 Jul;15(3):147-51. PMID 25202672
- [Background] Porcaro G, Brillo E, Giardina I, Di Iorio R. Alpha Lipoic Acid (ALA) effects on subchorionic hematoma: preliminary clinical results. Eur Rev Med Pharmacol Sci. 2015 Sep;19(18):3426-32. PMID 26439038
- [Derived] Costantino M, Guaraldi C, Costantino D. Resolution of subchorionic hematoma and symptoms of threatened miscarriage using vaginal alpha lipoic acid or progesterone: clinical evidences. Eur Rev Med Pharmacol Sci. 2016 Apr;20(8):1656-63. PMID 27160142